CLINICAL TRIAL: NCT05386849
Title: Demonstration of an Artificial Intelligence Based Closed Loop Glucose Control System as a Therapeutic Modality in Type 2 Diabetic Patients
Brief Title: Closed Loop Glucose Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ideal Medical Technologies (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IMT 2022-1
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Closed Loop Glucose Control; Artificial Pancreas; Artificial Intelligence; Glucose; Intensive Care Unit
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Early Feasibility Safety Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FUSION closed loop glucose control system (Experimental): All subjects will be treated with the FUSION closed loop glucose control system for up to 24 hours
  Interventions: Device: FUSION closed loop glucose control system

INTERVENTIONS:
Device: FUSION closed loop glucose control system — The FUSION system will be used to control the subjects glucose to a range of 100-140 mg/dL. Data will be collected for up to 24 hours, or upon early termination of the study session.

SUMMARY:
This is a proof of concept safety study of an artificial intelligence based closed loop glucose control system designed for use in the intensive care unit setting.

The type 2 diabetic subjects in this study will have their glucose controlled to a range of 100-140 mg/dL by a novel artificial intelligence based closed loop glucose control system for a period of 24 hours. The subjects will consume three standardized meals during the 24 hour study period.

DETAILED DESCRIPTION:
Tight glucose control in the intensive care unit (ICU) setting is difficult to achieve. The investigators hypothesize that a closed loop glucose control system based on artificial intelligence (AI) will improve upon the glucose control currently achieved by the current open loop manual methods, and that this improved glucose control may improve the outcomes of critically ill patients, including those with COVID-19.

This Earl Feasibility Study will test the ability of a prototype artificial intelligence based closed loop glucose control system named FUSION, to provide safe and effective glucose control in subjects with type 2 diabetes in a clinical research center (CRC) setting. Subjects with type 2 diabetes have been chosen as they are insulin resistant, which makes their insulin resistance profile similar to that of ICU patients. As this is the first in human study of a new medical device, the controlled environment of the CRC is preferable to the less controlled environment of an ICU setting.

The prototype FUSION system to be used in this study will consist to two Dexcom G6 continuous glucose monitors (CGM), the AI-based glucose control software run on an all-in-one medical computer, and two syringe pumps. The prototype system is housed on a medical cart. Based on the average glucose value of the two Dexcom G6 CGM's, and the rules of the FUSION systems AI-based glucose control software, the FUSION system will make rate adjustments every 5-10 minutes to the intravenous infusion rates of short acting insulin (NovoLog) and dextrose (D10NS) under its control, in an attempt to keep the subjects glucose in the range of 100-140 mg/dL. The FUSION system only requires entry of the subjects study identification number and weight in kilograms to initiate the system.

For safety reasons, the subjects will have their blood glucose independently measured every 10-60 minutes on a YSI 2900 glucose analyzer and the point of care Nova StatStrip system, throughout the 24 hour study period.

The study has halting criteria to avoid recurrent instances of severe hypoglycemia (< 54 mg/dL).

The average of the two CGM's, that is used by the FUSION system for glucose control, will be used for statistical analysis. In addition, both the average glucose value used by the FUSION system and each individual CGM system will be compared to the YSI glucose analyzer for correlation between systems using the Surveillance Error grid.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18-70 years of age, inclusive.
2. Can understand and sign an informed consent, communicate with the investigator, and understand and comply with the protocol requirements.
3. Have had a diagnosis of type 2 diabetes for a period of at least 3 months.
4. Use insulin injections at home for glucose control.
5. Have a hemoglobin A1c (HbA1c) in the range of 7.0 - 10.0%.
6. Have a hemoglobin in the normal range for sex:

   1. Females: 12-15.5 grams/dL.
   2. Males: 13.5-17.5 grams/dl.
7. Have adequate venous access sites in upper extremities.
8. Body weight between 40 - 150 kg.

Exclusion Criteria:

1. Have participated in an interventional medical, surgical, or pharmaceutical study within 30 days of screening.
2. Have a known hypersensitivity to any of the components of study treatment.
3. Have skin disease/injury at Dexcom G6 CGM insertion site(s) that would prevent insertion of the CGM.
4. Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion would cause the individual to be noncompliant.
5. Have a medical condition that in the opinion of the investigator could affect study participation and/or personal well-being.
6. Have a clinically significant history or presence of any of the following conditions:

   1. Hepatic failure or has alanine aminotransferase (ALT) greater than 3 times the upper limit of normal.
   2. Has an estimated GFR <30 ml/min/1.73 m2 or End Stage Kidney Disease on renal replacement therapy.
   3. Have congestive heart failure greater than class 1 on the NYHA classification system.
   4. Have a history of seizures.
   5. Have a history of cerebrovascular accident.
   6. Have a history of ischemic heart disease.
7. For female subjects of potential childbearing age (age 18 to 55) they will be excluded if:

   1. Pregnant.
   2. Refuse to agree to a pregnancy test at the time of enrollment.
   3. Have a positive urine pregnancy test at the time of enrollment.
8. Have a positive COVID-19 test within 14 days of visit 3.
9. Have any COVID-19 related symptoms in the 14-day period prior to visit 3.
10. Have a known unprotected COVID-19 exposure in the 14-day period prior to visit 3.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  The primary safety outcome will be the percent of all glucose values that are within the glucose range of less than 70 mg/dL.
Primary Efficacy Outcome | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  The primary efficacy outcome will be the percent of all glucose values that are within the glucose range of 70-180 mg/dL.

SECONDARY OUTCOMES:
Severe hypoglycemia | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  Measure the percent of all glucose values that are less than 54 mg/dL.
Hyperglycemia | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  Measure the percent of all glucose values that are greater than 180 mg/dL.
Glucose dispersion | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  Measure the degree of glucose dispersion by determining the coefficient of variation.
Time in desired control range | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  Measure the percent of all glucose values that are within the desired control range of 100-140 mg/dL.

OTHER OUTCOMES:
Average glucose value used by FUSION system versus from blood | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  The average glucose value used by the FUSION system in mg/dL will be compared with blood glucose in mg/dL from an arterialized hand vein. The arterialized hand vein measurement will occur every 10-60 minutes throughout the closed loop session.
Glucose readings from CGM's versus from blood | From beginning of use of the FUSION system to end of use of the FUSION system, which will be a period of time of up to 24 hours
  Glucose readings in mg/dL from the Dexcom G6 CGM's will be compared with blood glucose in mg/dL from an arterialized hand vein. The arterialized hand vein measurement will occur every 10-60 minutes throughout the closed loop session.

CONTACTS AND LOCATIONS:
Overall Officials: Leon DeJournett, MD, Study Director — Ideal Medical Technologies; Francisco Pasquel, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeJournett L, DeJournett J. In Silico Testing of an Artificial-Intelligence-Based Artificial Pancreas Designed for Use in the Intensive Care Unit Setting. J Diabetes Sci Technol. 2016 Nov 1;10(6):1360-1371. doi: 10.1177/1932296816653967. Print 2016 Nov. PMID 27301982
- [Background] DeJournett J, DeJournett L. Comparative Simulation Study of Glucose Control Methods Designed for Use in the Intensive Care Unit Setting via a Novel Controller Scoring Metric. J Diabetes Sci Technol. 2017 Nov;11(6):1207-1217. doi: 10.1177/1932296817711297. Epub 2017 Jun 22. PMID 28637358
- [Background] DeJournett J, Nekludov M, DeJournett L, Wallin M. Performance of a closed-loop glucose control system, comprising a continuous glucose monitoring system and an AI-based controller in swine during severe hypo- and hyperglycemic provocations. J Clin Monit Comput. 2021 Apr;35(2):317-325. doi: 10.1007/s10877-020-00474-2. Epub 2020 Jan 31. PMID 32006145
- [Background] DeJournett L. Essential elements of the native glucoregulatory system, which, if appreciated, may help improve the function of glucose controllers in the intensive care unit setting. J Diabetes Sci Technol. 2010 Jan 1;4(1):190-8. doi: 10.1177/193229681000400124. PMID 20167184
- [Background] Sardu C, D'Onofrio N, Balestrieri ML, Barbieri M, Rizzo MR, Messina V, Maggi P, Coppola N, Paolisso G, Marfella R. Outcomes in Patients With Hyperglycemia Affected by COVID-19: Can We Do More on Glycemic Control? Diabetes Care. 2020 Jul;43(7):1408-1415. doi: 10.2337/dc20-0723. Epub 2020 May 19. PMID 32430456